CLINICAL TRIAL: NCT07398742
Title: Incidence and Microbial Profiles of Periprosthetic Joint Infection After Total Knee Arthroplasty in Obese vs Non-Obese Patients
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Saber Muthanna Saber, Phd. student, Bispebjerg Hospital
Other Study IDs: p-2023-14433-Micro
Record Dates: First submitted 2025-09-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Knee Arthropathy; PJI
Keywords: microbiological profiles; knee arthroplasty; obesity; pji
MeSH Terms: conditions — Obesity; Juvenile polyposis syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with obesity: Patients with body mass index of 30 or more
- Patients without obesity: Patients with body mass index less than 30

SUMMARY:
Importance: After a primary total knee arthroplasty (TKA), we anticipate that obese individuals are more likely to experience a of periprosthetic joint infection (PJI). Knowing the microbial profile in obese patients can potentially help in choosing the proper prophylactic measures for this group as well as tailoring the empirical antibiotics in relation to PJI in obese patients.

Objective: To compare incidence of PJI revisions within 2 years after TKA in obese vs non-obese OA patients. Secondarily: To compare microbial profiles of infections in these groups in two time windows: early (≤90 days) vs late (91-730 days) and incidence of revisions due to all causes within 2 years.Design and Setting: We will include patients having primary knee arthroplasty using Danish national registers. Patients will be stratified into anthropometric groups, referred to as exposed and unexposed to obesity, based on their baseline Body Mass Index (BMI). Participants included in the analysis population will be followed up for 2 years, until first revision, death or migration whichever comes first.

Participants: We will include adult patients with available weight and height data with primary/idiopathic or secondary (due to meniscus or cruciate ligament lesion) OA who received primary TKA in the period from 2011-01-01 and 2021-02-28. Patients will be identified from the Danish knee arthroplasty register.

Exposure and Comparator: The cohort will be divided into obese (exposed), defined as body mass index (BMI) ≥ 30 kg/m2; and non-obese (unexposed), defined as BMI < 30 kg/m2.

Main Outcomes and Measures: The primary outcome will be revision due to prosthetic joint infection (PJI) within 730 days following TKA. Secondary endpoints will then be to examine revision due to all causes within 730 days following TKA and type of microbial infection between obese and non-obese in the first 90 days and the period from 91 days to 730 days following TKA.

Planned Statistical Analyses: We will use descriptive statistics to summarize the baseline characteristics of the two groups. Hazard ratios with corresponding two-sided 95% confidence intervals (95%CIs) for experiencing the outcome will be estimated using a Cox proportional hazards regression model. We will fit both unadjusted (crude) model and a propensity score adjusted model calculated based on age, sex, highest completed education, household income, comedications, and Elixhauser Comorbidity Measure (ECM), all collected up to the day of surgery. Stratified analyses will categorize PJI cases by bacterial infection and compare crude proportions between groups based on the absolute risk difference with 95% confidence intervals.

Ethical Considerations and Registration: The study and its statistical analysis plan will be registered in clinicaltrials.org prior to conducting the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults with available BMI data recieved knee arthroplasty due to osteoarthritis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to be eligible, we will include adult patients with primary or secondary osteoarthritis (due to meniscus or cruciate ligament lesion) who underwent primary TKA between January 1, 2011, and February 28, 2021, and for whom weight and height data are available. Patients will be identified from the DKR. Patients are followed for 2 years, until first revision, death or migration, whichever comes first.
Sampling Method: Non-Probability Sample
Enrollment: 101299 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Incidence Periprosthetic joint infection | 2 years
  PJI: our definition of PJI is adapted from The European Bone and Joint Infection Society (EBJIS) criteria as at least one of the following:
  A. Danish Knee Arthroplasty Register-registered revision surgery due to infection. B. At least 2 deep-tissue samples of phenotypically indistinguishable bacteria isolated from at least 3 deep-tissue samples C. One or more positive intraoperative samples from a closed fluid aspirate AND a biopsy (fluid AND tissue) of phenotypically indistinguishable bacteria isolated.

SECONDARY OUTCOMES:
Incidence of Revision due to all causes | 2 years
  Any registered surgery in the ipsilateral knee following the primary arthroplasty extracted from the danish knee arthroplasty register
Proportions Microbiological profiles in periprosthetic infection | 90 days
  For the revision due to PJI, we will stratify the outcome looking into the proportions of the following groups of bacteria A. PJI due to Staphylococcus aureus. B. PJI due to Coagulase-negative staphylococci. C. PJI due to other gram-positive bacteria. D. PJI due to gram-negative bacteria. E. PJI due to anaerobic bacteria. F. PJI due to mycoplasmic infection. G. PJI due to polymicrobial infection. H. PJI with negative culture.
Proportions of Microbiological profiles in periprosthetic infection | 91 days to 2 years
  For the revision due to PJI, we will stratify the outcome looking into the proportions of the following groups of bacteria A. PJI due to Staphylococcus aureus. B. PJI due to Coagulase-negative staphylococci. C. PJI due to other gram-positive bacteria. D. PJI due to gram-negative bacteria. E. PJI due to anaerobic bacteria. F. PJI due to mycoplasmic infection. G. PJI due to polymicrobial infection. H. PJI with negative culture.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedic surgery and traumatology, Bispebjerg Hospital, Copenhagen, Denmark, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT07398742/Prot_SAP_000.pdf